CLINICAL TRIAL: NCT02952612
Title: Active Surveillance of Papillary Thyroid Microcarcinoma (PTMC) in Catholic Medical Center
Brief Title: Active Surveillance of Papillary Thyroid Microcarcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dong Jun Lim (Other)
Responsible Party: Sponsor-Investigator, Dong Jun Lim, Professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Other Study IDs: KC16OISI0414
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Thyroid Cancer, Papillary
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Papillary thyroid microcarcinoma are small thyroid cancer measuring 1cm or less. Most of this tumor are not palpable and are identified either through pathologic examination or from imaging modalities, such as CT scan or thyroid sono. Active surveillance of papillary microcarcinoma is to observe thyroid papillary cancer without immediate surgical approach. The purpose of this study is to understand more about the characteristics of papillary microcarcinoma, which has been known for "the cancer slowly progression"

ELIGIBILITY:
Inclusion Criteria:

1. < 1 cm solitary nodule
2. Surrounded by ≥ 2 mm normal thyroid parenchyma
3. Subcapsular locations not adjacent to surrounding structures, recurrent laryngeal nerve, trachea, or carotid artery
4. No evidence of invasion to surrounding structures, recurrent laryngeal nerve, trachea or carotid artery
5. No extrathyroidal extension
6. Clinically N0 and Clinically M0
7. ≥ 18 years
8. Combined severe comorbidities or Inoperable condition (optional)
9. No wish to surgery and Willingness to accept active surveillance
10. No history of radiotherapy on head and neck area
11. Accepted by the Board of Thyroid Cancer Meeting

Exclusion Criteria:

1. ≥ 1 cm nodule and multifocal nodules regardless of size
2. Papillary thyroid carcinoma variants associated with poor prognosis (tall cell variant, columnar variant, hobnail variant) or other types of thyroid cancer)
3. Subcapsular locations adjacent to surrounding structures, recurrent laryngeal nerve, trachea or carotid artery
4. Evidence of invasion to surrounding structures, recurrent laryngeal nerve, trachea or carotid artery
5. Extrathyroidal extension
6. Any of N1 or M1
7. Documented increase in size according to America Thyroid Association (ATA) guideline in a previously confirmed Papillary thyroid microcarcinoma
8. < 18 years
9. Not willing to accept observational active surveillance approach

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This observational study enrolls patients who was diagnosed as papillary thyroid microcarcinoma by FNA (Fine needle aspiration) or CNA(Core needle aspiration) and who wish to be enrolled this study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Progression of papillary thyroid microcarcinoma | 5 years after enrollment
  Using thyroid sonography, check any changes in size and shape of papillary thyroid microcarcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Jun Lim, MD, PhD, Study Chair — Seoul St. Mary's Hospital
Locations (1):
- Seoul St Mary's Hospital, Seoul, Seocho-Gu, South Korea

IPD SHARING:
Plan to Share IPD: Yes